CLINICAL TRIAL: NCT05157711
Title: A Randomized, Placebo- and Benchmark-controlled, Double-blind Clinical Trial of Anusol Topical Ointment to Evaluate Symptom Relief in Patients With Haemorrhoids
Brief Title: Clinical Trial of Anusol Ointment for Symptom Relief in Patients With Haemorrhoids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST-20-U92
Record Dates: First submitted 2021-05-10; First posted 2021-12-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2021-11

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Zinc Oxide; bismuth subgallate; Peruvian balsam; bismuth oxide; Oxymetazoline; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anusol ointment (Experimental): Anusol ointment (Zinc oxide [10.75g], Bismuth subgallate [2.25 g], Balsam peru [1.875 g], Bismuth oxide [0.875 g] in each 100g of ointment).
  Interventions: Drug: Anusol
- Benchmark (Active Comparator): RELIEF® rectal ointment (phenylephrine hydrochloride 2.5mg/g), marketed
  Interventions: Drug: Relief [Name]
- Placebo (Placebo Comparator): Anusol ointment after the removal of the active ingredients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anusol — Daily at night and in the morning and after each bowel movement for two weeks
  Other Names: Anusol Ointment (Zinc oxide, Bismuth subgallate, Balsam peru), Bismuth oxide)
  Arms: Anusol ointment
Drug: Relief [Name] — Daily at night and in the morning and after each bowel movement for two weeks
  Other Names: RELIEF rectal ointment (phenylephrine hydrochloride)
  Arms: Benchmark
Drug: Placebo — Daily at night and in the morning and after each bowel movement for two weeks
  Other Names: Placebo ointment (Anusol ointment without active ingredients)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Anusol topical ointment for the relief of internal and external haemorrhoid symptoms in people with Grades I-III haemorrhoids compared to a placebo (the study medication without the active ingredients) and a benchmark product.

DETAILED DESCRIPTION:
Adult patients with haemorrhoids meeting all the eligibility criteria will be allocated in three study arms: test, placebo and benchmark. Approximately twenty-two subjects per group will be enrolled to assure that approximately 20 subjects in each group complete the study. The study will be conducted in Armenia.The study will last approximately 2 weeks for each subject and will consist of 3 visits. The first subject first visit is planned for June 2021, and the study will continue until the target sample size is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-75 years old.
2. Subjects with a diagnosis of symptomatic internal and/or external haemorrhoids, confirmed by Investigator as Grade I-III.*
3. Has at least two of the following haemorrhoid symptoms for at least two consecutive days immediately prior to screening: pain, discomfort, itching, irritation, burning, inflammation, swelling, bleeding, or defecation discomfort/difficulty.
4. Has at least two of the following haemorrhoid symptoms with at least moderate intensity (>4 reported by subject) at the baseline/screening: pain, discomfort, itching, irritation, burning, inflammation, swelling, bleeding or defecation discomfort/difficulty.
5. Non-pregnant, non-lactating female. Females should be able to distinguish rectal bleeding from menstrual vaginal bleeding.
6. In the case of a female of childbearing potential (CBP), using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device (IUD), condom with spermicide, diaphragm with spermicide, partner's vasectomy, bilateral tubal ligation). Abstinence or vasectomies are acceptable, but if the female subject's lifestyle or partner changes then she will agree to implement one of the other acceptable methods of birth control.
7. In the case of a female of child-bearing potential, has a negative urine pregnancy dipstick test (UPT) at Visit 1 prior to randomization and are willing to submit to a UPT at Visit 2 and at the end of study (EOS),
8. In the case of a female of non-childbearing potential, has had a hysterectomy or is postmenopausal (at least 1 year with no menses prior to enrollment).
9. Agrees not to participate in any clinical study from Visit 1 through end of study.
10. Read, understand and sign an informed consent.
11. Willing not to change their shampoo, soap or body washing products during the study.
12. Willing and able to comply with study instructions.

Exclusion Criteria:

1. Has anorectal condition(s) such as malignant tumors of the anus or rectum, fistula-in-ano or chronic sepsis, fissure-in-ano, incontinence, condylomata and Grade IV haemorrhoids.
2. History of previous proctological surgery.
3. Diagnosis of Inflammatory Bowel Disease (IBD).
4. Evidence or history of fecal incontinence.
5. Current diagnosis or history of an uncorrected coagulation defect or concurrently uses anticoagulants (except low dose aspirin or non-steroidals).
6. Is using medication which, in the opinion of the Investigator, will interfere with the study results.
7. Has known hypersensitivity or previous allergic reaction to any of the active or inactive components of the study products.
8. Use of stool softeners, but not on a stable regimen during the past 28 days prior to enrolling in the study.
9. Receiving treatment labeled or intended for haemorrhoids during the past 7 days prior to start of the study.
10. Receiving treatment labeled or intended for haemorrhoids throughout the study, other than the assigned product.
11. Use of local analgesics and/or anti-inflammatories during the past 14 days prior to the start of the study.
12. Receiving Monoamine oxidase inhibitors (MAOI) within the past 14 days prior to enrolling and during the study.
13. Has severe arterial hypertension, tachysystolic cardiac rhythm disturbance, decompensated heart failure, cardiac conduction disorders, severe hepatic failure, severe renal failure, thyrotoxicosis, acute pancreatitis, recurrent thromboembolism, granulocytopenia, or other clinically significant co-morbid condition, which, in PI's opinion, may affect the patient safety and/or affect participation in the study.
14. Female subjects who are lactating and/or pregnant or planning to become pregnant during the study.
15. Is currently participating in any clinical testing.
16. Has received any investigational drug(s) within 28 days before start of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Subject reported severity of heamorrhoid symptoms | Day 7
  Subject will grade severity of each hemorrhoid symptom (pain, itching, swelling, bleeding, discomfort, burning, inflammation, overall Irritation, defecation discomfort/difficulty) in 10 cm VAS, from 0 (None) to 10 (Most severe).
Subject reported severity of heamorrhoid symptoms | Day 14
  Subject will grade severity of each hemorrhoid symptom (pain, itching, swelling, bleeding, discomfort, burning, inflammation, overall Irritation, defecation discomfort/difficulty) in 10 cm VAS, from 0 (None) to 10 (Most severe).
Subject reported improvement of heamorrhoid symptoms | Day 7
  Subject will grade improvement of each haemorrhoid symptom (pain, itching, swelling, bleeding, discomfort, burning, inflammation, overall Irritation, defecation discomfort/difficulty) compared to Day 0 in 10 cm VAS from 0 (None) to 10 (Complete improvement).
Subject reported improvement of heamorrhoid symptoms | Day 14
  Subject will grade improvement of each haemorrhoid symptom (pain, itching, swelling, bleeding, discomfort, burning, inflammation, overall Irritation, defecation discomfort/difficulty) compared to Day 0 in 10 cm VAS from 0 (None) to 10 (Complete improvement).
Subject reported overall improvement of haemorrhoid symptoms | Day 7
  Subject will rate overall improvement of haemorrhoid symptoms compared to Day 0 in 10 cm VAS from 0 (None) to 10 (Complete Improvement).
Subject reported overall improvement of haemorrhoid symptoms | Day 14
  Subject will rate overall improvement of haemorrhoid symptoms compared to Day 0 in 10 cm VAS from 0 (None) to 10 (Complete Improvement).
Subject reported overall shrinkage of haemorrhoids | Day 7
  Subject will rate overall shrinkage of haemorrhoids compared to Day 0 in 10 cm VAS from 0 (None) to 10 (Complete Improvement).
Subject reported overall shrinkage of haemorrhoids | Day 14
  Subject will rate overall shrinkage of haemorrhoids compared to Day 0 in 10 cm VAS from 0 (None) to 10 (Complete Improvement).
Investigator reported severity of haemorrhoid symptoms and signs | Day 7
  Investigator will rate each haemorrhoid symptom and sign (erythema, swelling/edema, inflammation,dryness, overall irritation, haemorrhoid severity) in six-point scale from 0 (none) to 5 (very severe).
Investigator reported severity of haemorrhoid symptoms and signs | Day 14
  Investigator will rate each haemorrhoid symptom and sign (erythema, swelling/edema, inflammation,dryness, overall irritation, haemorrhoid severity) in six-point scale from 0 (none) to 5 (very severe).
Investigator reported overall improvement of haemorrhoid symptoms | Day 7
  Investigator will rate overall improvement of haemorrhoid symptoms compared to Day 0 in six-point scale from 0 (none) to 5 (complete improvement)
Investigator reported overall improvement of haemorrhoid symptoms | Day 14
  Investigator will rate overall improvement of haemorrhoid symptoms compared to Day 0 in six-point scale from 0 (none) to 5 (complete improvement)
Investigator reported overall shrinkage of haemorrhoids | Day 7
  Investigator will rate overall shrinkage of haemorrhoids compared to Day 0 in six-point scale from 0 (none) to 5 (complete improvement).
Investigator reported overall shrinkage of haemorrhoids | Day 14
  Investigator will rate overall shrinkage of haemorrhoids compared to Day 0 in six-point scale from 0 (none) to 5 (complete improvement).

OTHER OUTCOMES:
Overall product performance | Day 14
  Subjects who complete the study per protocol will complete an overall product performance questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Annahita Ghassemi, PhD, Study Director — Director, Global Product Safety & Clinical Affairs Church & Dwight Co., Inc.
Locations (2):
- Armenia (2):
  - Erebouni Medical Center, Yerevan
  - Izmirlyan Medical Center, Yerevan